CLINICAL TRIAL: NCT00983775
Title: Pharmacokinetic and Pharmacodynamic Profile of Rapid Acting Insulin Injected by Needle-free Jet-injection
Brief Title: Pharmacology of Insulin Injected With Jet-Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Cees Tack, MD PhD, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PKPD_SQ_1
Record Dates: First submitted 2009-09-21; First posted 2009-09-24 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Pharmacokinetic profile; Pharmacodynamic profile; insulin; jet injector
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- healthy low dose insulin (Experimental): 16 healthy non-diabetic volunteers. The type of insulin tested will be the rapid-acting insulin analogue insulin aspart (Novorapid®), at a dose of 0.2 units per kg body weight.
  Interventions: Device: jet injector (SQ pen/Novopen III)
- healthy high dose insulin (Experimental): 16 healthy non-diabetic volunteers. The type of insulin tested will be the rapid-acting insulin analogue insulin aspart (Novorapid®), at a dose of 0.4 units per kg body weight.
  Interventions: Device: jet injector (SQ pen/Novopen III)
- type 1 diabetes mellitus (Experimental): 16 people with type 1 diabetes mellitus. The type of insulin tested will be the rapid-acting insulin analogue insulin aspart (Novorapid®), at a dose of 0.4 units per kg body weight.
  Interventions: Device: jet injector (SQ pen/Novopen III)

INTERVENTIONS:
Device: jet injector (SQ pen/Novopen III) — The rapid-acting insulin analogue insulin aspart (Novorapid®), at a dose of 0.2 units per kg body weight, will be injected subcutaneously. On one experimental day insulin will be injected with the jet injector and placebo with the conventional insulin pen. On the other experimental day insulin will be injected with the conventional insulin pen and placebo with the jet injector.
  Other Names: SQ pen; Novopen III
  Arms: healthy low dose insulin
Device: jet injector (SQ pen/Novopen III) — The rapid-acting insulin analogue insulin aspart (Novorapid®), at a dose of 0.4 units per kg body weight, will be injected subcutaneously. On one experimental day insulin will be injected with the jet injector and placebo with the conventional insulin pen. On the other experimental day insulin will be injected with the conventional insulin pen and placebo with the jet injector.
  Other Names: SQ pen; Novopen III
  Arms: healthy high dose insulin; type 1 diabetes mellitus

SUMMARY:
The purpose of this study is to compare the pharmacological profile of insulin administered with jet-injection with that of insulin injected with a conventional insulin pen.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Body-mass index 18-28 kg/m2
* Blood pressure <160/90 mmHg
* Stable glycaemic control with HbA1c 6.5-9.0% (for patients with type 1 diabetes mellitus)
* Duration of diabetes >1 year (for patients with type 1 diabetes mellitus)

Exclusion Criteria:

* Inability to provide informed consent
* Chronic use of medication other than oral contraceptives or thyroid hormone replacement therapy (with stable euthyroidism for at least 3 months)
* Chronic use of medication other than insulin or low-dose angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) treatment (for patients with type 1 diabetes mellitus)
* Type 2 diabetes in first-degree relatives (for healthy subjects)
* History of a major cardiovascular disease event (myocardial infarction, stroke, symptomatic peripheral artery disease, coronary bypass surgery, percutaneous coronary or peripheral artery angioplasty)
* Pregnancy
* Macroalbuminuria, i.e. urinary albumin excretion >200 microg/min in collected urine sample or urinary albumin-to-creatinine ratio >300 mg/g in spot urine sample (for patients with type 1 diabetes mellitus)
* Symptomatic diabetic neuropathy (for patients with type 1 diabetes mellitus)
* Proliferative diabetic retinopathy (a history of proliferative retinopathy that was successfully treated with laser coagulopathy is not an exclusion criterion) (for patients with type 1 diabetes mellitus)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
(time to) maximal glucose infusion rate | 0-8 hours after insulin injection

SECONDARY OUTCOMES:
(time to) maximal insulin concentration | 0-8 hours after insulin injection

CONTACTS AND LOCATIONS:
Overall Officials: Cees J Tack, MD PhD, Study Chair — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, P.O. Box 9101, Netherlands